CLINICAL TRIAL: NCT02690766
Title: Translating Healthy Lifestyle Interventions for Breast and Endometrial Cancer Survivors With Diabetes
Brief Title: Translating Healthy Lifestyle Interventions for Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 15-0162; P30DK093002 (NIH)
Record Dates: First submitted 2016-02-18; First posted 2016-02-24 (Estimated); Last update posted 2023-05-16 (Actual); Status verified 2019-07

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent; Breast Cancer; Endometrial Cancer
Keywords: Cancer; Breast Cancer; Endometrial cancer,; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Breast Neoplasms; Endometrial Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Physical Activity Group (Other): The Success Study's Standard Behavioral Weight Change Intervention consists of 75 minute group sessions held monthly which include 30 minutes of physical activity with a licensed Physical Activity Instructor. Web Lessons that include information on Physical Activity, Nutrition and Healthy Behaviors will also be provided to participants on the study's website.
  Interventions: Behavioral: Standard Behavioral Weight Change Intervention

INTERVENTIONS:
Behavioral: Standard Behavioral Weight Change Intervention — Participants enrolled in Phase 2 of the study will meet once a month for 75 minutes over the course of 4 months. Within this 75 minutes, they will complete 25 minutes of physical activity with a licensed physical activity instructor that is very experienced with working with this population, review and discuss various topics/lessons that relate to diabetes, nutrition, survivorship and physical activity with the study's interventionist and Group Leader

SUMMARY:
Investigators proposed to refine and test the feasibility and acceptability of a 4-month multi-modal lifestyle intervention in African American female breast or endometrial cancer survivors diagnosed with type 2 diabetes.

DETAILED DESCRIPTION:
Recent systematic reviews and meta-analyses of cohort studies show that physical activity can reduce mortality and morbidity in diabetes and obesity-related cancers. Yet, there have been few efforts to promote physical activity within the context of female cancer survivorship, particularly among women with diabetes. In response, investigators proposed to refine and test the feasibility and acceptability of a 4-month multi-modal lifestyle intervention in African Americans (AA) with diabetes and who are breast or endometrial cancer survivors. This web-based, lifestyle intervention, coupled with coaching calls and in-person exercise sessions, may be an effective way to promote physical activity and healthy survivorship. The primary goal is for participants to participate in 30 minutes of moderate-to-vigorous physical activity five times a week. The investigators' aims : i) refine a theory-driven healthy lifestyle intervention, that is delivered via computer technologies and periodic in-person group exercise sessions with appropriate content, literacy demand and graphics, ii) assess the preliminary effects of the intervention on the primary outcome of level of moderate to vigorous physical activity (MVPA), as measured by accelerometry; weight, glycosylated hemaglobin and evaluate the effect of eating behaviors, wellbeing/functioning (quality of life, depressive symptoms, self-efficacy), compliance/adherence to protocol and acceptability on response to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* African American women, ages 30
* No evidence of pregnancy, as evidenced by negative urine pregnancy test.
* Diagnosed with type 2 diabetes by their provider
* Diagnosed with Stage I-III breast or endometrial cancer
* Completed treatment for breast or endometrial cancer at least 4 months and no more 5 years ago English-speaking
* Agree to participate in all aspects of the semi-structured interview (Aim 1)
* Agree to participate in all aspects of the feasibility study, including group sessions (Aim 2)
* Access to the internet via phone or computer
* Access to a working phone for personal use

Exclusion Criteria:

* Non-English speaking
* Recent epilepsy, cardiac event or stroke in last 6 months,special nutritional needs (e.g. current evidence of malignancy; HIV)
* History of epilepsy, cardiac event or stroke within the last year
* Known diagnosis of HIV
* Known new malignancy
* Less than 4 months or more than 2 years post treatment of Stage I-III breast or endometrial cancer.
* No diagnosis of type 2 diabetes
* No self-report of African American race/ethnicity
* No access to a phone for personal use
* No access to the internet via computer or mobile phone

Ages: 30 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in Body Weight | Week 0 and 16
  Body weight in pounds will be measured on a digital scale to assess change in body weight over the 16-week intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Wanda Nicholson, MD, Principal Investigator — University of North Carolina, Chapel Hill

IPD SHARING:
Plan to Share IPD: No